CLINICAL TRIAL: NCT05818358
Title: A Pilot Study to Examine the Effect of Consuming Beans and Whole Grains at Breakfast on Postprandial Vascular Responses in People With Arterial Stiffness
Brief Title: Postprandial Effects of Bean and Whole Grain Consumption on Arterial Stiffness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, Dr. Peter Zahradka, professor, University of Manitoba
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: HS25221
Record Dates: First submitted 2023-03-16; First posted 2023-04-18 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Arterial Stiffness

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Black Beans (cooked) (Active Comparator): At one of the three visits, participants will consume a ¾ cup of cooked black beans. Participants will be provided with 100 ml of water with the food, and will be allowed to drink up to another 150 mL of water during the 2 hour test period. The participants will not be blinded to the order and the type of food product they receive at a visit, however, the samples will be assigned a number to ensure the analytical team is blinded to the test product until the end of the study. Should the need to re-administer a test product arise, the participant will receive the test product from the same treatment number again at an extra visit after the original 3 visits have been completed.
  Interventions: Dietary Supplement: black beans
- Whole Wheat Grain (cooked) (Active Comparator): At one of the three visits, participants will consume a ¾ cup of cooked whole wheat grain. Participants will be provided with 100 ml of water with the food, and will be allowed to drink up to another 150 mL of water during the 2 hour test period. The participants will not be blinded to the order and the type of food product they receive at a visit, however, the samples will be assigned a number to ensure the analytical team is blinded to the test product until the end of the study. Should the need to re-administer a test product arise, the participant will receive the test product from the same treatment number again at an extra visit after the original 3 visits have been completed.
  Interventions: Dietary Supplement: wheat berries
- White Rice (cooked) (Placebo Comparator): At one of the three visits, participants will consume a ¾ cup of cooked white rice. Participants will be provided with 100 ml of water with the food, and will be allowed to drink up to another 150 mL of water during the 2 hour test period. The participants will not be blinded to the order and the type of food product they receive at a visit, however, the samples will be assigned a number to ensure the analytical team is blinded to the test product until the end of the study. Should the need to re-administer a test product arise, the participant will receive the test product from the same treatment number again at an extra visit after the original 3 visits have been completed.
  Interventions: Dietary Supplement: white rice

INTERVENTIONS:
Dietary Supplement: black beans — ¾ cup of cooked black beans
  Arms: Black Beans (cooked)
Dietary Supplement: wheat berries — ¾ cup of cooked whole wheat grain
  Arms: Whole Wheat Grain (cooked)
Dietary Supplement: white rice — ¾ cup of cooked white rice
  Arms: White Rice (cooked)

SUMMARY:
This is a single site, single-blinded, controlled randomized crossover clinical trial designed to compare the effects of black beans or whole grains or white rice at breakfast on postprandial vascular responses in males and females with arterial stiffness (n=10). Eligible participants will be asked to attend 3 in-person visits for comparative testing of black beans versus whole grains versus white rice.

DETAILED DESCRIPTION:
This is a single site, single-blinded, randomized, controlled crossover study designed to compare the vascular responses of males and females with arterial stiffness before and 2 hours after ingestion of black beans or whole grains (wheat) or white rice (isocaloric comparator).

Recruitment will consist of a total of 10 participants with arterial stiffness. Participants will be recruited through advertisement from the local community.

The study will be conducted at the Asper Clinical Research Institute, St. Boniface Hospital. Participants will be asked to provide written informed consent prior to participation in the study. Participants who have provided written consent will be asked to attend an in-patient screening visit to provide a fasting blood sample (and females a urine sample) and assess the presence of arterial stiffness (by PWV) to determine eligibility. Should the participant be eligible to participate, they will be scheduled for three study visits to obtain fasting blood samples and assess postprandial blood vessel function. During the first study visit period, participants will be asked to complete a Food Habits Questionnaire.

ELIGIBILITY:
Inclusion Criteria:

1. Male, or non-pregnant, non-lactating female, 45 to 65 years of age;
2. Brachial-ankle pulse wave velocity >1400 cm/s on at least one side;
3. Plasma creatinine ≤265 µmol/L;
4. Aspartate aminotransferase <160 U/L, andalanine aminotransferase <150 U/L;
5. Glycated hemoglobin ≤6.5%;
6. LDL-cholesterol <5 mmol/L;
7. Stable regime if taking vitamin and mineral/dietary/herbal supplements for the past 1 month and while participating in the study;
8. Has not donated blood or blood products (e.g. platelets) during the past 2 months and willing to continue doing so while participating in the study;
9. Not participating in another dietary intervention trial for the past month and willing to not start another dietary intervention trial for the duration of this study;
10. Willing to comply with the protocol requirements and procedures;
11. Willing to provide informed consent.

Exclusion Criteria:

1. Has experienced a cardiovascular event (e.g. heart attack, stroke) or had a surgical procedure for cardiovascular disease (e.g. bypass, stent), presence of clinically diagnosed cardiac arrhythmia or valve stenosis, chronic renal disease, liver disease (with exception of fatty liver), lung disease, rheumatoid arthritis, immune disorder or disease (e.g. multiple sclerosis, leukemia), cancer in the previous 5 years, neurological disorders, or gastrointestinal disorders;
2. Taking vasoactive medications (e.g., ACE inhibitors, ARBs, AGE-breakers, thiazolidinediones, beta-blockers, statins, insulin, etc.);
3. Blood pressure >160 mmHg systolic and/or >100 mmHg diastolic;
4. History of gastrointestinal reactions or allergies to beans, bean flour, wheat, wheat flour, gluten, or rice;
5. Body weight exceeds the capacity of the DEXA (350 lbs);
6. Current (within the past 30 days) bacterial, viral or fungal infection;
7. Bleeding disorder;
8. Amputations of upper or lower extremities on both sides;
9. Any acute medical condition or surgical intervention within the past 3 months;
10. Drug and/or alcohol abuse;
11. Psychological disorder(s);
12. Unable to fast overnight;
13. Unable to take prescribed medication without food;
14. Unable to obtain vascular function measurements and/or blood sample at the screening or first study visits;
15. Not fully vaccinated for COVID-19.

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-03-22 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline Augmentation index at 2 hours | Time points 0 (prior to consumption) and 2 hours post consumption.
  Pulse wave analysis using a SphygmoCor XCEL device will be used to measure the augmentation index (AIx), an indicator of arterial stiffness, prior to consumption of the test products, and at 2 hours post-consumption.
Change from baseline Reflection magnitude at 2 hours | Time points 0 (prior to consumption) and 2 hours post consumption.
  Pulse wave analysis using a SphygmoCor XCEL device will be used to measure the reflection magnitude, an indicator of arterial stiffness, prior to consumption of the test products, and at 2 hours post-consumption.

SECONDARY OUTCOMES:
Change from baseline blood pressure at 2 hours | Time points 0 (prior to consumption) and 2 hours post consumption.
  A SphygmoCor XCEL device will be used to measure the blood pressure prior to consumption of the test products, and at 2 hours post-consumption.

CONTACTS AND LOCATIONS:
Locations (1):
- Asper Clinical Research Institute, Winnipeg, Manitoba, Canada

REFERENCES:
- [Derived] Zahradka P, Perera D, Charney J, Taylor CG. Distinct Effects of Wheat and Black Bean Consumption on Postprandial Vascular Responses in People with Arterial Stiffness: A Pilot Randomized Cross-Over Study. Nutrients. 2025 Mar 27;17(7):1159. doi: 10.3390/nu17071159. PMID 40218917